CLINICAL TRIAL: NCT01913652
Title: Phase II Trial of Cabazitaxel in Metastatic or Inoperable Locally Advanced Dedifferentiated Liposarcoma
Brief Title: Ph II Cabazitaxel DD Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1202; 2012-003672-39 (EudraCT Number); cabazL06470 (Other: Sanofi)
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Dedifferentiated Liposarcoma
Keywords: dedifferentiated liposarcoma; cabazitaxel
MeSH Terms: conditions — Liposarcoma | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): INN: Cabazitaxel Cabazitaxel will be administered at a dose of 25 mg/m² by intravenous infusion, over 1 hour, on day 1 of each 21 day cycle.
  Treatment should be administered until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel
  Other Names: Jevtana

SUMMARY:
Soft tissue sarcomas (STS) are a rare group of malignant heterogenous tumors (> 50 histological subtypes, including liposarcoma, the commonest subtype of STS) with distinct genetic, pathological and clinical profiles, and varying patterns of tumor spread. The optimal cytotoxic treatment for this group of patients remains uncertain. Single agents which are most effective include doxorubicin and ifosfamide, but objective response rates and progression-free survival times remain modest. There is clearly a need to improve treatment options for liposarcoma. Eribulin, a antimicrotubule agent that targets the protein tubulin in cells, interfering with cancer cell division and growth , has demonstrated activity in STS. Therefore, it is reasonable to explore whether other anti-microtubule agent like cabazitaxel have a role in STS. Cabazitaxel has been shown to be a relatively safe, effective and tolerated. This drug has been approved by FDA for prostate cancer. The main objective of this trial is to determine whether cabazitaxel demonstrate sufficient antitumor activity for liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Local diagnosis of dedifferentiated liposarcoma
* Age 18-75 yrs
* WHO performance status 0-1
* Radiological or histological diagnosis of inoperable locally advanced or metastatic disease, with evidence of disease progression within the past 6 months
* Clinically and/or radiographically documented measurable disease within 21 days prior to randomization.At least one site of disease must be unidimensionally measurable according to RECIST 1.1.
* One previous chemotherapy regimen for locally advanced or metastatic dedifferentiated liposarcoma (this could include pre-operative chemotherapy for primary disease if subsequent complete resection was not achieved).
* Adequate haematological, renal and hepatic function
* Birth control measures
* Estimated life expectancy > 3 months
* Related adverse events from previous therapies ≤ Grade 1
* Written informed consent

Exclusion Criteria:

* More than 1 prior molecularly targeted therapy (e.g. CDK4 inhibitor). Any prior such therapy must be completed at least 4 weeks before randomization.
* Symptomatic CNS metastases
* Previous encephalopathy of any cause or other significant neurological condition
* Concurrent or planned treatment with strong inhibitors or inducers of cytochrome P450 3A4/5
* Pregnancy
* inflammation of the urinary bladder (cystitis)
* Other invasive malignancy within 5 years (exceptions of non-melanoma skin cancer, localized cervical cancer, localized and presumably cured prostate cancer or adequately treated basal or squamous cell skin carcinoma)
* Significant cardiac disease
* Uncontrolled severe illness or medical condition, other than DD liposarcoma
* Hypersensitivity to taxanes or their excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years from first patient in
  The primary endpoint will be progression free survival, assessed at 12 weeks after start of treatment

SECONDARY OUTCOMES:
Time to progression | 3 years from first patient in
Progression free survival | 3 years from first patient in
Overall survival | 3 years from first patient in
Objective tumor response | 3 years from first patient in
  Objective tumor response as defined by RECIST 1.1
Time to onset of response | 3 years from first patient in
  Time to onset of response will be measured for patients achieving an objective response
Duration of response | 3 years from first patient in
  Duration of response will be measured for patients achieving an objective response
Occurence of adverse events | 3 years from first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, for adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Hayward, MD, Principal Investigator — Western General Hospital, Edinburgh, United Kingdom
Locations (11):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen (117), Antwerp
  - Hopitaux Universitaires Bordet-Erasme - Institut Jules Bordet (101), Brussels
- France (3):
  - CHU de Dijon - Centre Georges-Francois-Leclerc (229), Dijon
  - Centre Leon Berard (227), Lyon
  - Assistance Publique - Hopitaux de Marseille - Hôpital de La Timone (287), Marseille
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori (704), Milan
  - Istituto Oncologico Veneto IRCCS - Ospedale Busonera (3908), Padua
- United Kingdom (4):
  - Clatterbridge Centre for Oncology NHS Trust - Clatterbridge Cancer Centre NHS Foundation Trust (659), Bebington
  - Western General Hospital, Edinburgh
  - Royal Marsden Hospital - Chelsea, London (613), London
  - The Christie NHS Foundation Trust (610), Manchester